CLINICAL TRIAL: NCT02517723
Title: A Randomized Controlled Clinical Trial (RCCT) to Test the Effectiveness of Narrative Exposure Therapy (NET) Versus Dialectical-Behavioral Therapy in Reducing Trauma Related Symptoms in Women Suffering From Borderline Personality Disorder (BPD) and Posttraumatic Stress Disorder (PTSD)
Brief Title: Narrative Exposure Therapy in Women With Borderline Personality Disorder and Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evangelisches Krankenhaus Bielefeld gGmbH (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Martin Driessen, Martin Driessen, Prof. Dr. med., Evangelisches Krankenhaus Bielefeld gGmbH
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NET_BPS+PTBS
Record Dates: First submitted 2014-01-06; First posted 2015-08-07 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Borderline Personality Disorder; Stress Disorders, Post-Traumatic
Keywords: Borderline Personality Disorder; comorbid Posttraumatic Stress Disorder; Narrative Exposure Therapy; Dialectical-Behavioral Therapy
MeSH Terms: conditions — Borderline Personality Disorder; Stress Disorders, Post-Traumatic | interventions — Dialectical Behavior Therapy; Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- SIC + NET (Experimental): Waiting List + Standard Inpatient Care + Narrative Exposure Therapy
  Interventions: Behavioral: Narrative Exposure Therapy; Behavioral: Standard Inpatient Care; Other: Waiting List
- SIC + DBT (Active Comparator): Waiting List + Standard Inpatient Care + Dialectical Behavior Therapy
  Interventions: Behavioral: Dialectical Behavior Therapy; Behavioral: Standard Inpatient Care; Other: Waiting List

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy — Narrative Exposure Therapy (NET) is based on Testimony Therapy in combination with cognitive behavioural exposure techniques and elements of client-centered counselling. The clients can restore their autobiographic memories about their traumatic experiences. In this way fragmentary memories are transformed into a coherent narrative structure. This practice enables the processing of painful emotions and the construction of clear contingencies of dangerous and safe conditions, generally leading to significant emotional recovery. Therapeutic aims are the reduction of PTSD-Symptomload via activation of fear-network and habituation of fear and the placement of traumatic experiences in a reconstructed, detailed and consistent autobiography.
  NET will be applied in eight sessions (90-120min/session) in a standardized, manualized manner.
  Other Names: NET
  Arms: SIC + NET
Behavioral: Dialectical Behavior Therapy — Dialectical behavior therapy is a cognitive behavioral treatment program developed by Marsha Linehan to treat suicidal clients meeting criteria for BPD. It directly targets suicidal behavior, behaviors that interfere with treatment delivery, and other dangerous, severe, or destabilizing behaviors.
  Via standard DBT patients improve behavioral capabilities, motivation for skillful behavior, generalization of gains to the natural environment, structuring the treatment environment so that it reinforces functional rather than dysfunctional behaviors. It also targets the therapist capabilities and motivation to treat patients effectively. Patients get weekly individual psychotherapy (1 h/wk), group skills training (3.75 h/wk), a weekly therapist consultation team meetings.
  Other Names: DBT
  Arms: SIC + DBT
Behavioral: Standard Inpatient Care — Unspecific group therapy that is identical in both groups (music therapy etc.)
  Other Names: SIC
Other: Waiting List — Treatment as usual in the community (no DBT, no exposure of trauma memories)

SUMMARY:
Narrative Exposure Therapy (NET) is an evidence-based trauma-focussed treatment, suitable for survivors of prolonged and repeated exposure to traumatic stress and childhood adversity. Patients with Borderline Personality Disorder (BPD) often suffer from a comorbid Posttraumatic Stress Disorder (PTSD) caused by multiple traumatic events. Therapeutic aims are the reduction of PTSD-Symptoms in these patients via activation of associative neural networks related to traumatic experiences and habituation of fear and the placement of traumatic experiences in a reconstructed, detailed and consistent autobiography. This practice enables the processing of and coping with painful memories and the construction of clear contingencies of dangerous and safe conditions, generally leading to significant emotional recovery. The investigators assume that using NET the reduction of PTSD symptom severity is greater compared to treatment by Dialectical-Behavioral Therapy (DBT).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* DSM-IV-TR diagnoses of BPD and PTSD
* legal competence
* none or stable medication
* illegal drug abstinence for at least the last 6 months
* capacity to consent and contract

Exclusion Criteria:

* other severe mental disorders (e.g., bipolar disorder, acute psychosis)
* simultaneous consumption of drugs
* simultaneous participation in other treatment-studies
* pregnancy or breastfeeding
* lack of capability to negotiate a no-suicide agreement
* suicide attempt or attempts during the 8 weeks prior to start of treatment
* perpetrator-contact
* Body Mass Index (BMI) < 16

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change from first investigation in Posttraumatic Symptom Severity at 18 months (Clinician-Administered PTSD Scale; CAPS) | first investigation (t1), after waiting list (3 months, t2), directly after therapy (3 months, t1), 1 year after therapy (15 months, t3)

SECONDARY OUTCOMES:
Change from first investigation in Borderline Symptome Severity at 18 months(Borderline Symptom Liste; BSL) | first investigation (t1), after waiting list (3 months, t2), directly after therapy (6 months, t3), 1 year after therapy (18 months, t4)
Change from first investigation in Severity of Dissociative Symptoms at 18 months (Fragebogen zu Dissoziativen Symptome ;FDS) | first investigation (t1), after waiting list (3 months, t2), directly after therapy (6 months, t3), 1 year after therapy (18 months, t4)
Change from first investigation in Severity of Depressive Symptoms at 18 months (Becks Depressions Inventar II, BDI-II) | first investigation (t1), after waiting list (3 months, t2), directly after therapy (6 months, t3), 1 year after therapy (18 months, t4)
Change from first investigation in Quality of Life at 12 months (WHO-Qualitiy of Life; WHOQOL) | first investigation (t1), after waiting list (3 months, t2), directly after therapy (6 months, t3), 1 year after therapy (18 months, t4)

CONTACTS AND LOCATIONS:
Overall Officials: Carolin Steuwe, M.Sc., Study Director — Clinic of Psychiatry, Evangelisches Krankenhaus Bielefeld; Martin Driessen, Prof. Dr. med., Principal Investigator — Clinic of Psychiatry, Evangelisches Krankenhaus Bielefeld
Locations (1):
- Clinic of Psychiatry, Evangelisches Krankenhaus Bielefeld, Bielefeld, Germany

REFERENCES:
- [Derived] Steuwe C, Berg M, Beblo T, Driessen M. Narrative Exposure Therapy in Patients With Posttraumatic Stress Disorder and Borderline Personality Disorder in a Naturalistic Residential Setting: A Randomized Controlled Trial. Front Psychiatry. 2021 Nov 26;12:765348. doi: 10.3389/fpsyt.2021.765348. eCollection 2021. PMID 34899426
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Steuwe C, Rullkotter N, Ertl V, Berg M, Neuner F, Beblo T, Driessen M. Effectiveness and feasibility of Narrative Exposure Therapy (NET) in patients with borderline personality disorder and posttraumatic stress disorder - a pilot study. BMC Psychiatry. 2016 Jul 20;16:254. doi: 10.1186/s12888-016-0969-4. PMID 27439618